CLINICAL TRIAL: NCT03123640
Title: Improving Drug Safety in Emergency Patients -a Randomized Controlled Trial
Acronym: EPIMERR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diakonhjemmet Hospital (Other)
Collaborators: Diakonhjemmet Hospital Pharmacy (Unknown); Diakonhjemmet Foundation (Unknown); University of Oslo (Other)
Responsible Party: Principal Investigator, Lisbeth Damlien Nymoen, Ph.d. candidate and project pharmacist, Diakonhjemmet Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: EPIMERR -2015/1356/REK sør-øst
Record Dates: First submitted 2017-04-12; First posted 2017-04-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Medication Compliance; Drug-Related Side Effects and Adverse Reactions; Remission; Medicinal Substance; Adverse Effect; Drug Interaction Potentiation
Keywords: Medication reconciliation; Medication review; Drug related admission
MeSH Terms: conditions — Medication Adherence; Drug-Related Side Effects and Adverse Reactions | interventions — Medication Reconciliation; Medication Review

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial With intervention Group and Control group
Masking Description: Not possible to mask the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Pharmacist conducts medication reconciliation and medication review while the patient is admitted to the emergency Department. The pharmacist present results from medication reconciliation to physicians at the emergency Department before the Medical history is obtained. Further the pharmacist will discuss drug related problems obtained during the medication review with the physicians to customize and optimize the medication treatment for each patient.
  Interventions: Other: Medication reconciliation and medication review
- Control group (No Intervention): Standard treatment without pharmacist intervention in the emergency department

INTERVENTIONS:
Other: Medication reconciliation and medication review — Pharmacist performed medication reconciliation and medication review
  Arms: Intervention group

SUMMARY:
Aim/Objective: Investigate the effect of implementing a working model for performing medication reconciliation (MR) and medication review (MRe) in the emergency department (ED), on readmissions, patient safety and efficiency of the stay in the ED and the hospital. Research design: randomized, controlled, non-blinded trial. Control group; standard care. Intervention group; MR and MRe performed at admission to the ED by a clinical pharmacist in the interdisciplinary team. The intervention is based on a working model for MR, developed in our initiation project, and it will be adapted to also include MRe. Key challenges in this research field: Currently no implemented systematic model ensuring that the patient's correct medication list is obtained and assessed at the point of admission. There is lack of studies investigating the clinically outcome of performing MR and MRe in the ED. Lack of knowledge on the extent of drug related hospital admissions in Norway. These challenges are also recognized and prioritized by the Norwegian authorities. Impact and utility: The results from this study will give important answers to the challenges listed above. The results could imply a huge impact on how to organize ED in Norway regarding drug safety. If the hypothesis of this study is confirmed, implementing the intervention described will increase patient safety, both the hospital and society can reduce health care expenses from readmissions, and also the readmission-burden can be reduced for the patients.

DETAILED DESCRIPTION:
Inclusion and randomization procedures

Staff at the emergency department, including physicians and nurses will be informed about the project. At admission, the project pharmacist will describe the project to each potential participant and/or their next of kin, then provide written information about the project and answer potential questions. If patients temporary are unable to consent when asked to participate (e.g. delirium) their next of kin will be asked to supply a preliminary consent in the patients place. If the patient later refuses to participate he/she will be excluded from the trial, and any registered data for this patient will be deleted. Patients will periodically be included at day shift and evening shift and by different clinical pharmacists to reduce potential bias. We will randomize the patients into two study groups. The randomization process will be conducted by Department of Biostatistics and Epidemiology at Oslo University Hospital. This department will deliver randomization lists, and the project pharmacist will follow randomization procedure.

Data registration

Patient data will be registered on paper forms, which will be de-identified after the patient data is transferred de-identified to the password protected project database on the hospital research server. Only a code list will connect the patient to his or her data. Paper forms will at all times be kept accessible only to authorized project personnel, and eventually the forms will be maculated. De-identified patient information will not be brought out of the hospital. The code list connecting the patients to their data will at the latest be deleted 3 years after start of data collection. When results are published it will not be possible to identify individual patients.

Customized Standard Operating Procedures addressing inclusion and randomization operations, registry operations and how to perform the intervention is developed.

Sample size calculation

Available information about readmission frequency at Diakonhjemmet Hospital is based on 30 days follow-up, and therefore cannot be used to calculate proportion of patients readmitted after 12 months. However, numbers from Oslo University Hospital estimate a readmission proportion of 50% after 12 months in a comparable patient population. Therefore this estimate is used as the expected readmission rate in the control group of this project. In a previous Swedish study conducted by Ulrika Gillespie who is member of the reference group of this project, a 16% reduction in hospital revisits within 12 months was found amongst older patients (>80 years) following a comparable intervention as described in this project. On this basis, it will be necessary to include at least 146 patients in each group to show a significant effect on the primary endpoint (significance level of 5%, study power of 80%). However, the elderly patients included in the Swedish study had more comorbidity and therefore more use of health care resources. In this project we will include all patients 18 years and older and thereby the difference between the control group and intervention group probably will be smaller. A more realistic difference between the groups is 10%; thereby 385 patients would have to be included in each group to show a significant effect on the primary endpoint. To compensate for dropout the aim is to include 400 patients in each project group, thus a total of 800 patients. Based on statistics from Diakonhjemmet Hospital, inclusion of this amount of patients from the Emergency Department would require an inclusion period of 12 months.

Statistics and analysis

Statistical analyses will be conducted in IBM (International Business Machines)SPSS Statistics (Statistical Package for the Social Sciences). Data will be assessed for normality and analyzed according to appropriate statistical tests. The baseline demographic and clinical characteristics will be summarized using proportions, means and standard deviations, or median and interquartile range, as appropriate. Baseline comparisons: Characteristics of project participants in the two project groups will be compared using the chi-square test for categorical variables and the Student's t-test or non-parametric equivalent (e.g. the Mann-Whitney U test) for continuous variables. Multivariable analysis (logistic regression) will be used to compare endpoints between project groups while adjusting for prognostic variables and potential confounders. All statistical tests will be interpreted with a significance level of 5% (two-tailed). For building the model for prioritizing patients at increased risk of drug-related admissions and drug-related problems at admission to the emergency department binary regression analysis will be used. Data will be analyzed according to intention-to-treat (ITT) principles. In addition to ITT analysis, per protocol analysis will also be performed.

Approval

The project is approved by the Regional committee for medical and health research ethics (REC) and the research committee at Diakonhjemmet Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years admitted to the emergency department
* Able and willing to provide written consent (see Inclusion and randomization procedures and 6.Ethics)

Exclusion Criteria:

* Patient have previously been included
* Terminal ill patients with short life expectancy
* Control group patients where physician at the emergency department request an assessment from a clinical pharmacist
* Control group patients where the project pharmacist reveal drug-related problems of major clinical relevance and has to intervene

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 806 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2018-05-16 (Actual); Study Completion 2022-09-04 (Actual)

PRIMARY OUTCOMES:
Proportion of patients readmitted | 12 months from inclusion
  Difference between intervention- and control group in proportion of patients readmitted

SECONDARY OUTCOMES:
Proportion of patients readmitted | 6 months from inclusion
  Difference between intervention- and control group in proportion of patients readmitted
Average number of admissions | 12 months from inclusion
  Difference between intervention- and control group in average number of admissions
Time to next contact with a hospital | Time to next readmission, maximum 12 months from inclusion
  Difference between intervention- and control group in time to next contact with a hospital
Proportion of patients not hospitalized following admission to the emergency department (patients which condition is resolved in the emergency department) | During the relevant hospital admission (at inclusion)
  Difference between intervention- and control group in proportion of patients not hospitalized following admission to the emergency department
Length of stay at the emergency department | During the relevant hospital admission (at inclusion)
  Difference between intervention- and control group in length of stay at the emergency department
Overall length of hospital stay | During the relevant hospital admission (at inclusion)
  Difference between intervention- and control group in overall length of hospital stay
Investigate the efficiency of the new working model (for conducting medication reconciliation and medication review) | During inclusion period
  Use a semi structural questionnaire to investigate the efficiency of the new working model
Identify risk factors correlated to medication related admissions and drug related problems | Retrospective, 18 months after inclusion start (24. April 2017)
  Identify risk factors correlated to medication related admissions and drug related problems and use binary regression to build a prioritizing model, evaluate and test the model
High risk patients | Retrospective, 18 months after inclusion start (24. April 2017)
  Compare high risk patients for medication related admissions and drug related problems to high risk patients for clinical relevant medication discrepancies
Drug related admission | By pharmacist during the relevant hospital admission (at inclusion), by physicians and multidisciplinary team; retrospective, 18 months after inclusion start (24. April 2017)
  Describe the frequency of drug related admissions in the intervention group, and describe consequences, out-come and follow-up for these patients.
Patients point of view | 2 years after inclusion start (24. April 2017)
  To reveal the patients point of view for adjustment of the intervention: Describe patients view on medication regimen, believes and concerns about medication, medication lists and drug-related admissions using results from group interview and survey amongst a randomized sample of patients. 10% of the included patient will retrospectively be invited to participate in the group interview and 25% of the included patient will retrospectively be invited to fill out a survey
Retrospectively testing the two prioritizing models | Retrospective, 2 years after inclusion start (24. April 2017)
  To investigate the effect our two prioritizing models can have on patient safety we will retrospectively investigate the proportion of high risk patients for clinical relevant medication discrepancies and high risk patients for medication related admissions, for those readmitted in the control group and the intervention group.

CONTACTS AND LOCATIONS:
Overall Officials: Erik H Øie, PhD, MD, Study Chair — Diakonhjemmet Hospital
Locations (1):
- Diakonhjemmet Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nymoen LD, Flatebo TE, Moger TA, Oie E, Molden E, Viktil KK. Impact of systematic medication review in emergency department on patients' post-discharge outcomes-A randomized controlled clinical trial. PLoS One. 2022 Sep 19;17(9):e0274907. doi: 10.1371/journal.pone.0274907. eCollection 2022. PMID 36121830